CLINICAL TRIAL: NCT02505191
Title: A Pilot Phase I, Randomised, Open Mono-center, Multiple Dose, Two Parallel Groups Clinical Trial Investigating the Pharmacokinetics of a Prolonged-release Formulation in Comparison to an Immediate-release Formulation of St. John's Wort Extract Ze 117 in Healthy Male Volunteers Under Fasting Condition
Brief Title: Pilot Pharmacokinetic Study of a Prolonged-release Formulation of St. John's Wort Extract Ze 117
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Max Zeller Soehne AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ze117-1-2014-01a
Record Dates: First submitted 2015-06-22; First posted 2015-07-22 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Pharmacokinetics
MeSH Terms: interventions — Delayed-Action Preparations; Hypericum extract LI 160

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test (Experimental): St. John's wort prolonged-release tablet 500 mg
  Interventions: Drug: St. John's wort prolonged-release tablet 500 mg
- Reference (Active Comparator): St. John's wort film coated tablets 250 mg (Remotiv N)
  Interventions: Drug: St. John's wort film coated tablets 250 mg

INTERVENTIONS:
Drug: St. John's wort prolonged-release tablet 500 mg
  Other Names: Prolonged-release formulation
  Arms: Test
Drug: St. John's wort film coated tablets 250 mg
  Other Names: Immediate-release formulation
  Arms: Reference

SUMMARY:
A pilot phase I, randomised, open mono-center, two parallel group clinical trial investigating the pharmacokinetics of a prolonged-release formulation in comparison to an immediate-release formulation of St. John's wort extract Ze 117 in healthy male volunteers under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian male volunteers
* Physically and mentally healthy as judged by means of a medical and standard laboratory examination
* BMI of between 19 and 29 kg/m2, inclusively
* Weight not exceeding 90 kg
* Non-smokers (confirmed by urine cotinine test)
* Informed cConsent as documented by signature

Exclusion Criteria:

* Known or suspected hypersensitivity to any ingredient of the investigational medicinal product
* Any clinically significant illnesses or clinically significant surgery within 1 year prior to the administration of the study medication
* Any surgical or medical condition which might interfere with absorption, distribution, metabolism or excretion of the drug
* Any clinically significant abnormality or abnormal laboratory test results, as judged by the investigator found during the medical screening
* Positive test of hepatitis B, hepatitis C or HIV screening (HIV antibody, Hepatitis B (HBsAg), Hepatitis C (HCV)
* ECG abnormalities (clinical significant) or vital signs abnormalities (systolic blood pressure lower than 90 or over 145 mmHg, diastolic blood pressure lower than 60 or over 95 mmHg, or heart rate less than 45 or over 100bpm) at screening
* History of asthma or obstructive pulmonary disease (e.g.COPD)
* Known photohypersensitivity.
* Presents or history of alcohol dependence within the last year (> 40 g ethanol/d or more than 10 units per weeks (1unit=150 ml of wine or 360 ml of beer or 45 ml alcohol 45%))
* History of drug dependence or positive results of drug screen
* Concomitant participation in another clinical trial within the 4 weeks prior to the planned first drug administration.
* Donation of blood or blood products within 30 days prior to the planned first drug administration.
* Treatment with any medication or topical drugs with systemic action used in the past 4 weeks, prior to the planned first drug administration ,or 6 times the half-life of the respective drug, whatever is longer (excluding single use of paracetamol or ibuprofen up to 24 hours prior to the planned first drug administration).
* Suspected inability, e.g. language problems, or known or suspected non-compliance, e.g. non-willingness to fulfil the dietary restrictions
* Difficulty to swallow study medication
* Enrolment of the investigator, his/her family members, employees and other dependent persons
* Any reason which, in the opinion of the Investigator, would prevent the subject from participating the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Half Value Duration (HVD) of surrogate markers of the total extract Ze 117 | 3 days

SECONDARY OUTCOMES:
Peak-trough fluctuation (PTF) of surrogate markers of the total extract Ze 117 | 3 days
Tmax of surrogate markers of the total extract Ze 117 | 3 days
AUCss of surrogate markers of the total extract Ze 117 | 3 days
Cmax of surrogate markers of the total extract Ze 117 | 3 days
Cmin of surrogate markers of the total extract Ze 117 | 3 days
lag time of surrogate markers of the total extract Ze 117 | 3 days
Mean Residence Time (MRT) of surrogate markers of the total extract Ze 117 | 3 days
T1/2 of surrogate markers of the total extract Ze 117 | 3 days
Half value Duration (HVD) of hyperforin | 3 days

OTHER OUTCOMES:
Number of Adverse Events as a Measure of Safety and Tolerability | 7 days
  Physical examinations, Vital signs, 12 lead ECG, Clinical chemistry Parameters, Adverse Events records

CONTACTS AND LOCATIONS:
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany